CLINICAL TRIAL: NCT05677815
Title: The Effect of COVID-19 Infection on Post-operative Complications in Patients Underwent Surgery During the COVID-19 to Lift the Lockdown in China: Cohort Stdy
Brief Title: The Effect of COVID-19 Infection on Post-operative Complications
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Other Study IDs: KY20232002
Record Dates: First submitted 2023-01-08; First posted 2023-01-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Surgery; Postoperative Complications
Keywords: COVID-19; Postoperative Complications; Surgery
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with COVID-19 infection underwent surgery in 2023: Surgery was defined as any procedure done by a surgeon in an operating theatre under general, regional
  Interventions: Procedure: Underwent Surgery from 2019 to 2022
- patients without COVID-19 infection underwent surgery in 2023: Surgery was defined as any procedure done by a surgeon in an operating theatre under general, regional
  Interventions: Procedure: Underwent Surgery from 2019 to 2022

INTERVENTIONS:
Procedure: Underwent Surgery from 2019 to 2022 — Surgery was defined as any procedure done by a surgeon in an operating theatre under general, regional, or local anaesthesia

SUMMARY:
We did an multi-centre, observational cohort study in patients who had surgery in 2023. We included participants who underwent surgery after the COVID-19 to lift the lockdown in China. Patients meeting the same criteria were eligible who had been treated during the same calendar period of 2019 through 2021. The primary outcomes were the post-operative in-hospital complications. We hypothesized that the post-operative in-hospital complications during the COVID-19 to lift the lockdown period in China were different to complications for the same kind of patients during the same calendar period of the previous years.

DETAILED DESCRIPTION:
The outbreak of COVID-19 and its global pandemic have posed a threat to public health. The deadly virus, SARS-CoV-2, has been evolving to new, more infectious variant and other lineages with additional immune escape mutations. The highly transmissible Omicron variant has been present for around one year and has supplanted Delta as the leading strain in the global pandemic. Despite the fact that 656 million people have been infected with SARS-CoV-2 worldwide as of January 1, 2023, asymptomatic infections and mild cases account for more than 90% because of its notably declined pathogenicity.As of December 20, 2022, more than 130 sub-branches of Omicron have been imported into China, with BA.5.2 and BF.7 being the most prevalent strains.

On December 7, 2022, the State Council of China issued an announcement on further optimization of measures for preventing and controlling the COVID-19 epidemic ( easing of rigorous "zero COVID" policies). Since then, the rapid spread of COVID-19 has caused a surge of COVID-19 infections in the majority of China. As of January 6, a total of 503302 individuals have been infected. Consequently, the proportion of surgical patients with current or previous SARS-CoV-2 infections will inevitably increase within a short period of time. It has been reported that recovery from SARS-CoV-2 infection is associated with a transiently elevated risk of postoperative complications. The longer the time interval between SARS-CoV-2 infection and surgery, the lower the risk of postoperative complications. An updated recommendation suggested postponing surgery for at least seven weeks following SARS-CoV-2 infection, thereby reducing the risk of postoperative complications and 30-day mortality to baseline levels (similar risk with patients without a history of SARS-CoV-2 infection). However, these recommendations were based on limited data from the earlier Covid-19 pandemic (mostly caused by the Delta strain) in Europe and the United States It may not be feasible to generalize and apply this experience and consensus to the Chinese population and use it to guide current practice.

In this prospective cohort study, the postoperative complications will be described and compared in patients with or without Covid-19 infection. In addition, risk factors in the patients and surgical levels that are associated with an increase in postoperative morbidities and mortalities will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Underwent surgery at Xijing Hospital after the COVID-19 to lift the lockdown in China, effective as of 29th December in 2022 to 7th January in 2023.

Exclusion Criteria:

* Patients who had missing primary information data (i.e., postoperative information).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The exposure of interest was a diagnosis of COVID-19 viral infection defined using the the process of experiencing typical COVID-19 symptoms, or swab-test positive (either PCR or rapid antigen SARS-CoV-2 test). Patients with COVID-19 were categorised as symptomatic if they had concomitant respiratory illness or indicating respiratory support.
Sampling Method: Non-Probability Sample
Enrollment: 3350 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | postoperative in-hospital or 7-day complication
  Any postoperative in-hospital or 7-day complications, were based on the Clavien-Dindo Classified, and more than 0 grade was defined as complication.

SECONDARY OUTCOMES:
Severe post-complications | postoperative in-hospital or 7-day complication
  The complications classified greater than Clavien-Dindo II were defined as severe; ie, any complications that led to a reintervention (III), a life-threatening organ dysfunction (IV), or death (V).
in-hospital mortality | postoperative in-hospital or 7-day complication
  The proportion of patients who died during hospitalization post-operatively.
Critical care admission | postoperative in-hospital or 7-day complication
  The proportion of patients who admitted to ICU post-operatively.
Duration post-operative hospital stay | postoperative in-hospital or 7-day complication
  The time from end of operation to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang L, Zheng Z, Zhu S, Luo G, Gao B, Ma Y, Xu S, Dong H, Lei C. Changes in early postoperative outcomes and complications observed in a single center during the 2022 COVID-19 pandemic wave in China: A single-center ambispective cohort study. Chin Med J (Engl). 2023 Jul 20;136(14):1708-1718. doi: 10.1097/CM9.0000000000002724. Epub 2023 Jun 15. PMID 37310058
- [Derived] Zheng Z, Gao B, Luo G, Wang L, Lei C. Impact of SARS-CoV-2 infection on postoperative complications of patients undergoing surgery after general outbreak in China: a protocol for multicentre prospective cohort study. BMJ Open. 2023 Aug 24;13(8):e072608. doi: 10.1136/bmjopen-2023-072608. PMID 37620255